CLINICAL TRIAL: NCT04816331
Title: Follow-up of Inflammatory Responses and Multiorgan Outcomes FoLlowing Neonatal Brain injurY
Acronym: FIREFLY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Prof. Eleanor Molloy, Professor of Paediatrics & Child Health, Paediatrics, University of Dublin, Trinity College
Other Study IDs: ILP-POR-2019-086
Record Dates: First submitted 2021-03-02; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Neonatal Encephalopathy
Keywords: Brain Injuries; Multiple Organ Failure; Infant; Inflammation; Neutrophils
MeSH Terms: conditions — Brain Injuries; Multiple Organ Failure; Inflammation | interventions — Medical Records; Surveys and Questionnaires; Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Peripheral venous samples Urine Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonatal Encephalopathy (NE): This study is a follow up of children at 2-3 years of age who were enrolled in the HRB-funded Neonatal Inflammation and Multiorgan dysfunction and Brain injUry reSearch group (NIMBUS) project. These babies had Neonatal Encephalopathy and required Therapeutic Hypothermia and are matched with controls. Detailed antenatal, birth, resuscitation, oxygen requirements throughout inpatient stay and detailed neonatal intensive care management were collected. In addition, details of Therapeutic Hypothermia treatment including initiation, duration and clinical examination, investigations including cranial USS, MRI, EEG and placental histology analysis performed as were recorded.
  Interventions: Other: Medical records and clinical measurements
- Controls: The controls include age-matched normal children born at term with a normal delivery and postnatal course.
  Interventions: Other: Medical records and clinical measurements

INTERVENTIONS:
Other: Medical records and clinical measurements — Medical records and clinical measurements: Detailed antenatal, birth, resuscitation, oxygen requirements throughout inpatient stay and detailed neonatal intensive care management will be collected. Therapeutic Hypothermia treatment including initiation, duration and clinical examination, and investigations such as scans. In addition, clinical data will include medication, neurological (paediatric developmental psychologist assessment and Bayley Scales of Infant and Toddler Development) and multiorgan examination.
  Questionnaires for caregivers to assess social-emotional and adaptive domains.
  Tissue samples analysis and processing: Samples of blood, urine and saliva will be used for laboratory testing.
  Biomarker correlation with Multiorgan outcomes using statistical analysis: Data collected from medical records, clinical measurements, questionnaires, and tissue processing will be analysed using SPSS software for statistical analysis and modelling.
  Other Names: Questionnaires for caregivers to assess social-emotional and adaptive domains; Tissue samples analysis and processing: blood, saliva and urine

SUMMARY:
Babies who have brain injury also frequently have involvement of their kidneys, lung and heart. Although clinical care in the neonatal period is well defined there are few guidelines and evidence for developmental, heart and kidney followup in childhood. The investigators aim to develop and implement guidelines for health care workers and families on Followup after Neonatal Brain Injury.

Inflammation is an important factor in brain injury of newborns and also affects their heart lungs and other parts of their body. The investigators will use tests from the newborn period to predict outcome and help parents with planning health needs for their baby rather than waiting until any issues arise later on. By understanding inflammation the investigators can find methods to decrease the negative effects and improve outcomes in the future for babies and families.

DETAILED DESCRIPTION:
Neonatal brain injury is an important cause of neonatal death and disability such as cerebral palsy. Perinatal global hypoxic ischemic associated with Neonatal Encephalopathy (NE) results in multi-organ dysfunction which may persist in later childhood. In addition perinatal inflammation has been associated with neonatal brain injury and implicated in adult neuropsychiatric conditions.

The investigators aim to examine multi-organ dysfunction in early childhood in children who had NE by examining detailed cardiac, renal, neurological, haematological and neurodevelopmental outcomes. The investigators have previously defined detailed multi organ dysfunction (MOD) in this cohort in the neonatal period in infants with NE including organ outcomes as well as serum, urine and cerebrospinal fluid (CSF) biomarkers. They are now age-appropriate for detailed neurocognitive assessment and correlation with these biomarkers and the investigators plan to compare with age- matched controls. Immunological markers such as the inflammasome and microRNAs are altered in the neonatal period and may persist in early childhood. The investigators will modify negative inflammatory responses in vitro with specific antagonists as well as correlating these immune biomarkers with outcomes.

Quantifying multiorgan dysfunction in the neonatal period to ensure appropriate follow-up of all organs is merited. This would help in advanced clinical planning and long term follow up. In addition, understanding, the immune response in these children with NE and exploring systemic inflammation holds promise for future development of immunomodulatory adjunctive therapies and biomarkers to predict outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children at 2-3 years
* With diagnosis of Neonatal Encephalopathy
* Required Therapeutic Hypothermia

Exclusion Criteria:

-

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children at 2-3 years of age who were enrolled in the HRB-funded Neonatal Inflammation and Multiorgan dysfunction and Brain injUry reSearch group (NIMBUS) project. These babies had Neonatal Encephalopathy and required Therapeutic Hypothermia and are matched with controls.
  Patients recruited as part of the NIMBUS study in 3 Dublin Maternity Hospitals: the National Maternity hospital (NMH), the Rotunda hospital & the Coombe Women's and Infant's University Hospital (CWIUH) with an average of 120 infants with Neonatal encephalopathy (NE) Grade I-III deliveries per annum. This study will enrol 100 infants with NE and 100 controls (recruited in Tallaght University Hospital). The controls include age-matched normal children born at term with a normal delivery and postnatal course.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cardiovascular dysfunction in childhood | Children at 2-3 years of age
  It will be determined by normal or abnormal echocardiography using Tissue doppler and functional imaging.
Number of participants with renal dysfunction in childhood | Children at 2-3 years of age
  It will be assessed using renal scoring systems such as the Kidney disease Improving Global Outcomes (KDIGO) Acute Kidney injury score (scores 1 to 3, being 3 worse outcome) and measuring the concentration of urinary biomarkers (in mg/L) such as albumin, B2 microglobulin, Cystatin c, EGF, NGAL, OPN and UMOD. Deviations of the reference range values for the scores and urinary biomarkers will indicate renal dysfunction. Results will be reported as number of patients with renal dysfunction in childhood.
Number of participants with haematological anomalies persisting in childhood | Children at 2-3 years of age
  Number of patients with signs of coagulopathy will be defined using three indicators: APTT/PT (units per seconds), fibrinogen (mg/dL) and Leukocyte/neutrophil (percentage and units per Liter). Deviations of the reference range values for the three indicators will point to haematological anomalies. Results will be reported as number of patients with signs of coagulopathy.
Number of participants with neurological outcomes | Children at 2-3 years of age
  Presence or absence of seizures, motor and sensory dysfunction will be evaluated using Serial Cranial ultrasounds.

SECONDARY OUTCOMES:
Number and identity of miRNAs upregulated or downregulated in blood of participants. | Children at 2-3 years of age
  Between 350 and 800 miRNAs will be assessed in serum from patients and controls.
Fold change of inflammasome components (NLRP3 and ASC) in RNA isolated from blood of participants. | Children at 2-3 years of age
  Using RNA extracted from whole blood of patients and controls, the fold change RNA expression of inflammasome components (NLRP3 and ASC) will be evaluated.
Concentration level in pg/mL of multicytokines in serum of participants. | Children at 2-3 years of age
  Multiplex cytokine analysis will be performed and reported in pg/mL in serum. Cytokines to be included: Interleukin-1 alpha (IL-1α), Interleukin-1 beta (IL- 1β), Interleukin-6 (IL-6), Interleukin-8 (IL-8), Interleukin-10 (IL-10), Tumour Necrosis Factor-alpha (TNF-α), Interferon-gamma (IFN-δ), Vascular Endothelial Growth Factor (VEGF), Granulocyte Colony Stimulating Factor (G-CSF) and Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF), Erythropoietin, Neuronal glial fibrillary acidic protein (GFAP), ubiquitin carboxyl-terminal hydrolase L1 and S100B.
Bayley Scales of Infant and Toddler development (BSID III) scores of participants. | Children at 2-3 years of age
  Bayley Scales of Infant and Toddler development (BSID III) score is an assessment instrument designed to measure motor, cognitive, language, social-emotional, and adaptive behavior development in babies and young children. Composite scores are derived for cognitive, language, and motor development and scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160. Scores lower than 85 indicating mild impairment, and lower than 70 indicating moderate or severe impairment. Scores equal or higher than 85 indicate normal development.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Molloy, Prof., Principal Investigator — Professor of Paediatrics & Child Health, Paediatrics
Locations (5):
- Ireland (5):
  - The Coombe Women & Infants University Hospital, Dublin
  - The National Maternity Hospital, or Holles Street Hospital, Dublin
  - The Rotunda Hospital, Dublin
  - The Tallaght University Hospital, Dublin
  - Trinity College Dublin, The University of Dublin, Dublin

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be process within the research team associated to the project as per Ethical agreement with the corresponding ethical committees and explicit consent with parents/guardians of the patients.

REFERENCES:
- [Background] Aslam S, Molloy EJ. Biomarkers of multiorgan injury in neonatal encephalopathy. Biomark Med. 2015;9(3):267-75. doi: 10.2217/bmm.14.116. PMID 25731212
- [Background] Murray DM, O'Connor CM, Ryan CA, Korotchikova I, Boylan GB. Early EEG Grade and Outcome at 5 Years After Mild Neonatal Hypoxic Ischemic Encephalopathy. Pediatrics. 2016 Oct;138(4):e20160659. doi: 10.1542/peds.2016-0659. Epub 2016 Sep 20. PMID 27650049
- [Background] Chalak LF, Nguyen KA, Prempunpong C, Heyne R, Thayyil S, Shankaran S, Laptook AR, Rollins N, Pappas A, Koclas L, Shah B, Montaldo P, Techasaensiri B, Sanchez PJ, Sant'Anna G. Prospective research in infants with mild encephalopathy identified in the first six hours of life: neurodevelopmental outcomes at 18-22 months. Pediatr Res. 2018 Dec;84(6):861-868. doi: 10.1038/s41390-018-0174-x. Epub 2018 Sep 13. PMID 30250303
- [Background] Armstrong K, Franklin O, Sweetman D, Molloy EJ. Cardiovascular dysfunction in infants with neonatal encephalopathy. Arch Dis Child. 2012 Apr;97(4):372-5. doi: 10.1136/adc.2011.214205. Epub 2011 Jul 27. PMID 21798875
- [Background] Kirkley MJ, Boohaker L, Griffin R, Soranno DE, Gien J, Askenazi D, Gist KM; Neonatal Kidney Collaborative (NKC). Acute kidney injury in neonatal encephalopathy: an evaluation of the AWAKEN database. Pediatr Nephrol. 2019 Jan;34(1):169-176. doi: 10.1007/s00467-018-4068-2. Epub 2018 Aug 28. PMID 30155763
- [Background] Morkos AA, Hopper AO, Deming DD, Yellon SM, Wycliffe N, Ashwal S, Sowers LC, Peverini RL, Angeles DM. Elevated total peripheral leukocyte count may identify risk for neurological disability in asphyxiated term neonates. J Perinatol. 2007 Jun;27(6):365-70. doi: 10.1038/sj.jp.7211750. Epub 2007 Apr 19. PMID 17443199
- [Background] Buck BH, Liebeskind DS, Saver JL, Bang OY, Yun SW, Starkman S, Ali LK, Kim D, Villablanca JP, Salamon N, Razinia T, Ovbiagele B. Early neutrophilia is associated with volume of ischemic tissue in acute stroke. Stroke. 2008 Feb;39(2):355-60. doi: 10.1161/STROKEAHA.107.490128. Epub 2007 Dec 27. PMID 18162626
- [Background] Dammann O, Durum S, Leviton A. Do white cells matter in white matter damage? Trends Neurosci. 2001 Jun;24(6):320-4. doi: 10.1016/s0166-2236(00)01811-7. PMID 11356502
- [Background] Jenkins DD, Rollins LG, Perkel JK, Wagner CL, Katikaneni LP, Bass WT, Kaufman DA, Horgan MJ, Languani S, Givelichian L, Sankaran K, Yager JY, Martin RH. Serum cytokines in a clinical trial of hypothermia for neonatal hypoxic-ischemic encephalopathy. J Cereb Blood Flow Metab. 2012 Oct;32(10):1888-96. doi: 10.1038/jcbfm.2012.83. Epub 2012 Jul 18. PMID 22805873
- [Background] O'Hare FM, Watson RW, O'Neill A, Segurado R, Sweetman D, Downey P, Mooney E, Murphy J, Donoghue V, Molloy EJ. Serial cytokine alterations and abnormal neuroimaging in newborn infants with encephalopathy. Acta Paediatr. 2017 Apr;106(4):561-567. doi: 10.1111/apa.13745. Epub 2017 Feb 16. PMID 28097694
- [Background] O'Hare FM, Watson RW, O'Neill A, Blanco A, Donoghue V, Molloy EJ. Persistent systemic monocyte and neutrophil activation in neonatal encephalopathy. J Matern Fetal Neonatal Med. 2016;29(4):582-9. doi: 10.3109/14767058.2015.1012060. Epub 2015 Feb 19. PMID 25694256
- [Background] Lin CY, Chang YC, Wang ST, Lee TY, Lin CF, Huang CC. Altered inflammatory responses in preterm children with cerebral palsy. Ann Neurol. 2010 Aug;68(2):204-12. doi: 10.1002/ana.22049. PMID 20695013
- [Background] Hedtjarn M, Mallard C, Iwakura Y, Hagberg H. Combined deficiency of IL-1beta18, but not IL-1alphabeta, reduces susceptibility to hypoxia-ischemia in the immature brain. Dev Neurosci. 2005 Mar-Aug;27(2-4):143-8. doi: 10.1159/000085986. PMID 16046848
- [Background] Chevin M, Guiraut C, Sebire G. Effect of hypothermia on interleukin-1 receptor antagonist pharmacodynamics in inflammatory-sensitized hypoxic-ischemic encephalopathy of term newborns. J Neuroinflammation. 2018 Jul 30;15(1):214. doi: 10.1186/s12974-018-1258-6. PMID 30060742
- [Background] Ozaki E, Campbell M, Doyle SL. Targeting the NLRP3 inflammasome in chronic inflammatory diseases: current perspectives. J Inflamm Res. 2015 Jan 16;8:15-27. doi: 10.2147/JIR.S51250. eCollection 2015. PMID 25653548
- [Background] Looney AM, O'Sullivan MP, Ahearne CE, Finder M, Felderhoff-Mueser U, Boylan GB, Hallberg B, Murray DM. Altered Expression of Umbilical Cord Blood Levels of miR-181b and Its Downstream Target mUCH-L1 in Infants with Moderate and Severe Neonatal Hypoxic-Ischaemic Encephalopathy. Mol Neurobiol. 2019 May;56(5):3657-3663. doi: 10.1007/s12035-018-1321-4. Epub 2018 Sep 3. PMID 30178296
- [Background] Yang Z, Zhong L, Xian R, Yuan B. MicroRNA-223 regulates inflammation and brain injury via feedback to NLRP3 inflammasome after intracerebral hemorrhage. Mol Immunol. 2015 Jun;65(2):267-76. doi: 10.1016/j.molimm.2014.12.018. Epub 2015 Feb 21. PMID 25710917
- [Background] Fleiss B, Gressens P. Tertiary mechanisms of brain damage: a new hope for treatment of cerebral palsy? Lancet Neurol. 2012 Jun;11(6):556-66. doi: 10.1016/S1474-4422(12)70058-3. Epub 2012 May 16. PMID 22608669
- [Background] Sweetman DU, Onwuneme C, Watson WR, Murphy JF, Molloy EJ. Perinatal Asphyxia and Erythropoietin and VEGF: Serial Serum and Cerebrospinal Fluid Responses. Neonatology. 2017;111(3):253-259. doi: 10.1159/000448702. Epub 2016 Dec 1. PMID 27902983
- [Background] Eliwan HO, Watson RW, Aslam S, Regan I, Philbin B, O'Hare FM, O'Neill A, Preston R, Blanco A, Grant T, Nolan B, Smith O, Molloy EJ. Neonatal brain injury and systemic inflammation: modulation by activated protein C ex vivo. Clin Exp Immunol. 2015 Mar;179(3):477-84. doi: 10.1111/cei.12453. PMID 25204207
- [Background] Sarnat HB, Sarnat MS. Neonatal encephalopathy following fetal distress. A clinical and electroencephalographic study. Arch Neurol. 1976 Oct;33(10):696-705. doi: 10.1001/archneur.1976.00500100030012. PMID 987769
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Singh Y, Roehr CC, Tissot C, Rogerson S, Gupta S, Bohlin K, Breindahl M, El-Khuffash A, de Boode WP; European Special Interest Group 'Neonatologist Performed Echocardiography' (NPE). Education, training, and accreditation of Neonatologist Performed Echocardiography in Europe-framework for practice. Pediatr Res. 2018 Jul;84(Suppl 1):13-17. doi: 10.1038/s41390-018-0078-9. PMID 30072809
- [Background] Barkovich AJ, Hajnal BL, Vigneron D, Sola A, Partridge JC, Allen F, Ferriero DM. Prediction of neuromotor outcome in perinatal asphyxia: evaluation of MR scoring systems. AJNR Am J Neuroradiol. 1998 Jan;19(1):143-9. PMID 9432172
- [Background] Lawn JE, Lee AC, Kinney M, Sibley L, Carlo WA, Paul VK, Pattinson R, Darmstadt GL. Two million intrapartum-related stillbirths and neonatal deaths: where, why, and what can be done? Int J Gynaecol Obstet. 2009 Oct;107 Suppl 1:S5-18, S19. doi: 10.1016/j.ijgo.2009.07.016. PMID 19815202